CLINICAL TRIAL: NCT06162884
Title: Imaging Signature of Progressive Pulmonary Fibrosis in Idiopathic Pulmonary Fibrosis and Non-IPF Interstitial Lung Diseases
Brief Title: Single Time Point Prediction as Earlier Diagnosis of Progressive Pulmonary Fibrosis
Acronym: IS-PPF
Status: Recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Grace Hyun Kim, Principal Investigator, University of California, Los Angeles
Other Study IDs: IRB#23-001246; ECR2022-3630 (Other Grant/Funding Number: US Boehringer Ingelheim Pharmaceuticals, Inc.)
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Fibrosis
Keywords: imaging outcome; Single Timepoint Prediction; AI/machine learning; progressive ILD
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Medical imaging CT images will divide two arms of high STP and low STP groups using a threshold of 30% STP score.
  Blood collection: CPT, EDTA, Blood RNA and SST Nasal Swab: 2 nasal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- STP >=30%: STP score is 30% or greater than 30% in whole lung at baseline inspirational HRCT scan. STP score is an AL/ML derived score using radiomic patterns of lung parenchyma to identify the spatial location of likely progressed in the short-term follow up. The higher score is the worse expected outcome.
- STP < 30%: STP score is less than 30% in whole lung at baseline inspirational HRCT scan.

SUMMARY:
This study is a prospective observational study for subjects with idiopathic pulmonary fibrosis (IPF) or non-IPF interstitial lung diseases (ILD).

The purpose of this study is to compare whether imaging patterns from high-resolution computed tomography (HRCT) at baseline can predict worsening. Single Time point Prediction (STP) is a score derived from an artificial intelligenc/ machine learning (AI/ML) using the radiomic features from a HRCT scan that quantifies the imaging patterns of short-term predictive worsening.

DETAILED DESCRIPTION:
Primary objective is to predict early for progression in both IPF and non-IPF ILD population using an artificial intelligence (AI)/Machine Learning (ML) algorithm of STP score. The primary interest is to validate STP score in identifying a cohort early for the candidate of anti-fibrotic treatment. The study plans to collect clinical information such as pulmonary function tests (PFT), symptom scores, 6-minute walk tests (6MWT), and radiologic information from HRCT. This study does not intervene with patient's standard medical care.

This proposal is a prospective study that will enroll patients from the UCLA ILD Center. STP scores of subjects' baseline HRCT images will be grouped to one of 2 arms based on the baseline HRCT.

* Arm A: STP>=30% in whole lung
* Arm B: STP < 30% in whole lung

A subject's allocation will be determined by the baseline HRCT scan. STP score will be derived from the baseline HRCT to compare the early prediction of progression in ILD, STP of 30% threshold is expected to be close to the mean of overall population. In addition, a multi-scale guided attention (MSGA) is an imaging marker from deep learning model with two attention models to classify an IPF-likeliness using HRCT.

Primary endpoint of progression-free survival (PFS) is uniformly defined in IPF and non-IPD ILD subjects by the reduction of 10% or more by FVC in volume or 15% or more by DLCO or death from any cause, whichever came first.

Key secondary endpoint of this study are:

In IPF, progression-free survival (PFS) is defined by the reduction of 10% or more by FVC in volume or 15% or more by DLCO or death from any cause, whichever came first.

In non-IPF ILD, PFS is defined by two worsening outcomes out of three elements of PFT worsening, radiological worsening or symptom or disease-related death alone.

* Worsening in PFT is defined by 5% or more absolute decreases in the percent predicted FVC or 10% or more absolute decrease in the percent predicted DLCO.
* Radiological evidence of disease progression is defined by visual worsening (one or more of the following) from a radiological report or quantitative lung fibrosis (QLF) changes >=2% in whole lung
* Symptomatic worsening can be measure by King's Brief Interstitial Lung Disease (K-BILD) or Leicester Cough Questionnaire (LCD).

Secondary outcomes of this study are:

* To compare additional PFS criteria between two arms of STP
* To compare overall survival between the two arms of STP
* To compare the changes in 6-minute walk tests between the two arms of STP
* To compare PFS between two groups of MSGA marker positive and negative
* To compare overall survival between two groups of MSGA marker positive and negative

With a chronic ILD or IPF, lung function may be stable for a few years or continue to deteriorate slowly or rapidly develop more scar tissues over time. While it is known that age, biological sex, and lung function are factors that can impact risk of worsening lung function, there is a great need for better methods to predict which patients are at risk of worsening lung function. Having better methods to predict disease progression could allow more timely treatment with anti-fibrotic treatment to prevent the disease progression.

In both IPF and non-IPF ILD, HRCT scan is required for diagnosis. Imaging patterns derived from HRCT, called STP is designed to predict the areas in lung that may be likely to progress in the next 6 to 12 months. High STP scores are associated with poor prognosis and worsening the pulmonary function. The goal of this study is to test whether an AI-algorithm, the STP score from a single CT study, can predict disease progression in subjects with IPF and non IPF-ILD in a prospective study. This AI-algorithm was developed under NIH-sponsored study.

The purpose of prospective observational cohort study from UCLA is to test for the early sign of progressive fibrosis using baseline HRCT. This study, Imaging Signature of Progressive Pulmonary Fibrosis (IS-PPF) Research is a prospective study that will collect information regarding HRCT images, pulmonary function test, 6-minute walk, symptomatic score, and patients' clinical information to set up AI-driven imaging signature for evaluating the STP in predicting progression in IPF and non-IPF ILD.

This is an observational study; only minimally invasive procedures will be performed with study subjects (blood draws and nasal swabs). These biological samples will support future research studies. The study subject's will participation in the study for up to 3 years, the length of participation may vary. All subjects will continue to receive their usual care and treatment.

In summary, this research will create an opportunity to test and validate the imaging score and early prediction for IPF and non-IPF ILD that can impact current and future care practices.

ELIGIBILITY:
IPF Inclusion Criteria:

* Established a diagnosis (within 5 years) of IPF by enrolling center as defined by ATS/ERS/JRS/ALAT criteria
* Age over or equal to 40 years old
* No history of lung transplant
* FVC % predicted >= 45%
* DLCO % predicted >=25%
* Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control. WOCBP taking oral contraceptives (OCs) also have to use one barrier method.

Non-IPF ILD Inclusion Criteria:

* Established a diagnosis (within 5 years) of non-IPF ILD by enrolling center.
* Age over or equal to 18 years old
* Presence of chronic fibrosis ILD defined as architectural distortions with reticulation and the presence of traction bronchiectasis estimating visually >5% in whole lung.
* Patients treated with immunosuppressive agents (other than corticosteroids) for an underlying systemic disease need to be on a stable treatment for at least 12 weeks prior to screening
* FVC % predicted >= 45%
* DLCO % predicted >=25%
* Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control. WOCBP taking oral contraceptives (OCs) also have to use one barrier method

Exclusion Criteria:

* Planned to participate in an intervention trial within the next 6 months
* Currently listed for lung transplantation at the time of enrollment
* Malignancy, treated or untreated, other than malignancy unlikely to affect prognosis in the next 3 years such as skin cancer or non-metastatic prostate cancer within the past 5 years
* Any clinically significant co-morbidity, which in the view of investigator, is likely to contribute to mortality or ability to perform PFT's in the next 2 years
* Prebronchodilator Forced Expiratory Volume in 1 second (FEV1)/Forced vital capacity (FVC) <0.7 at as screening
* Exclusion of co-morbidities: congestive heart failure (stroke, deep vein thrombosis, pulmonary embolism, myocardial infarction), current virus-associated community acquired pneumonia, smoking-related chronic obstructive lung disease with FEV1 <70%, history of lung cancer, history of other cancer treated within the past 4 years for IPF and 5 years for non-IPF ILD (excluding basal cell carcinoma of skin).

HRCT data from subjects with combined pulmonary fibrosis and emphysema (CPFE) can be collected.

Major Discontinuing Criteria in this study

* lung transplant after baseline or death
* withdraw of consent or transition to another care center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary objective is to predict early for progression in both IPF and non-IPF ILD population using a new artificial intelligence machine learning (AI/ML) algorithm of Single Timepoint Prediction (STP) score from HRCT.
  The primary interest is to validate STP score in identifying cohort early for the candidate of anti-fibrotic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-11-22 (Estimated); Study Completion 2028-08-19 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) between the two arms by Single Time point Prediction (STP) score | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  PFS of IPF and non-IPF ILD will be compared in patients with STP >=30% or <30%. A higher STP score, ranging from 0% to 100%, indicates a worse outcome. Progression is uniformly defined in both IPF and non-IPF ILD population as the reduction of FVC >=10% or the reduction of DLCO >=15% or death due to the disease.

SECONDARY OUTCOMES:
Progression Free Survival (PFS2-PFS5) between the two arms by Single Time point Prediction (STP) score | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  Four additional PFS definitions will be used to test STP >=30% or <30%.
  * Key Secondary PFS definition (PFS2): same PFS in the primary endpoint for IPF or PPF definition for non-IPF (two events out of three elements in PFT (reduction of 5% or more in % predicted FVC or 10% or more in predicted DLCO if available; radiological worsening; symptomatic worsening);
  * Secondary PFS definition (PFS3) I: Key Secondary PFS definition (PFS2) convention for non-IPF or annual QLF increase of 2% or higher or visual worsening for IPF;
  * Secondary PFS definition (PFS4) II: Secondary PFS3 or 6 min walk (decrease of > 25m in the 6-minute walk distance) or QoL (KBILD of 4-point increase or LCQ SGRQ of 310-point reduction) for both IPF and non-IPF;
  * Secondary PFS definition (PFS5) III: Secondary PFS 4 or new Oxygen usage or increase in Oxygen usage (>1L of O2 per min) for both IPF and non-IPF
Overall Survival (OS) between the two arms by Single Time point Prediction (STP) score | From date of randomization until the date of death from any cause, assessed up to 3 years.
  Overall Survival will be compared with STP >=30% or <30%.
Changes in Distance Walked (Meters, m) on the 6-Minute Walk Test (6MWT) by two arms of STP score | From Baseline in every 3-6-month to end of the study (up to 2 years)
  The 6MWT measures the distance a patient is able to walk quickly on a flat, hard surface in a period of 6 minutes. The 6MW can ranges from 0 m to 1000m. In healthy subjects, the 6MWT ranges from 400m to 700m.
PFS between two arms by Multi-Scale Guided Attention (MSGA) marker | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Progression Free Survival will be compared in subjects with MSGA positive or negative marker.
OS between two arms by Multi-Scale Guided Attention (MSGA) marker | From Baseline to end of the study (up to 3 years)
  Overall Survival of IPF and non-IPF ILD will be compared in patients with MSGA positive or negative marker.

OTHER OUTCOMES:
Nasal and Blood Biobanking | At baseline (or screening) and year 1 follow-up
  The biorepository of nasal and blood samples will be collected for future ancillary study proposal.
Estimate median PFS by the levels of STP ranging 20% to 50% | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Progression Free Survival of IPF and non-IPF ILD will be compared in patients with a various threshold of STP 20% to 50%

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Weigt, MD, Principal Investigator — UCLA Division of Pulmonary, Critical Care, and Hospitals; Jonathan Goldin, MD, Principal Investigator — Radiological Sciences at the University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided